CLINICAL TRIAL: NCT04371705
Title: Efficacy of Ultrasound Guided Erector Spinae Plane Block in Patients Undergoning Abdominal Surgery
Brief Title: Efficacy of Ultrasound Guided Erector Spinae Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hassan Mokhtar Elshorbagy Hetta, assistant lecturarl, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Efficacy of ESPB
Record Dates: First submitted 2020-04-27; First posted 2020-05-01 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Hemodynamic Instability; Patient Satisfaction; Postoperative Pain; Regional Block
Keywords: ESPB; postoperative pain; Regional block
MeSH Terms: conditions — Patient Satisfaction; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESPB group (Experimental): 31 patients Will undergo ultrasound guided ESP block with 40 ml bupivacaine 0.25% (20 ml on each side).
  Interventions: Procedure: Erector spinae plane block
- control group (Placebo Comparator): 31 patients anesthetized with the protocol followed by Minia University Hospital
  Interventions: Other: control

INTERVENTIONS:
Procedure: Erector spinae plane block — The ESP block will be performed into a fascial plane between the deep surface of erector spinae muscle and the transverse processes using ultrasound guide.
  Arms: ESPB group
Other: control — placebo
  Arms: control group

SUMMARY:
Thoracic epidural and paravertebral blocks are the most widely regional technique used for postoperative analgesia after surgery, but they are difficult to perform and carry a risk of serious complication. In this study, investigator asses the efficacy of ultrasound ESPB on intraoperative and postoperative hemodynamics and patient satisfaction

DETAILED DESCRIPTION:
This prospective, double-blinded, randomized, controlled study was conducted at the period from October 2018 to December 2019. Sixty adults' patients ASA I-III, their ages ranged from 25-60 years undergoing abdominal surgery under general anesthesia. Each patient assigned written informed consent before the block performance.

Patients refused, known allergy to the used drugs, with history of coagulopathy, major organ failure and obesity (BMI>40 kg/m2) were excluded from the study.

Patients were randomly allocated into two equal groups by a computerized randomization table: ESPB group, and control group. The patient and the staff providing the postoperative care were blinded to the group assignment.

ESPB group: Will undergo ESP block with 40 ml bupivacaine 0.25% (20 ml on each side) control group: anesthetized with the protocol followed by Minia University Hospital.

Anesthetic technique was standardized for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age18-70 .
2. Both gender.

4. ASA I-III .

Exclusion Criteria:

1. patient refuse
2. Drug allergy.
3. Morbid obesity (BMI >40 kg/m2).
4. Psychiatric disorder.
5. Opioid dependence .

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Total Fentanyl Requirement | 24 hours
  The total amount of postoperative fentanyl in milligram

SECONDARY OUTCOMES:
Time of First Post Operative Analgesic Request | 24 hours
  the pain will be assisted based on the time for the first dose of rescue analgesia.
heart rate (HR) | 24 hours
  Hemodynamic
mean arterial pressure (MAP ) | 24 hours
  Hemodynamic

CONTACTS AND LOCATIONS:
Overall Officials: Nagy S. Ali, MD, Study Chair — Minia University Hospital
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No